CLINICAL TRIAL: NCT06937996
Title: Outcomes of Ablation of Unresectable Pancreatic Cancer Using the NanoKnife Irreversible Electroporation (IRE) System
Brief Title: Outcomes of Ablation of Unresectable Pancreatic Cancer Using the NanoKnife Irreversible Electroporation System-
Status: Recruiting | Type: Observational
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: E-24-987
Record Dates: First submitted 2025-04-11; First posted 2025-04-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer Non-resectable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: NanoKnife — The NanoKnife, System has been commercially available since 2009, and is FDA-approved to treat soft tissue tumors. The NanoKnife System has received FDA clearance for the surgical ablation of soft tissue. It has not received clearance for the therapy or treatment of any specific disease or condition.

SUMMARY:
The purpose of this study is to evaluate the short and intermediate term safety of the NanoKnife Irreversible Electroporation System when used off-label to treat unresectable pancreatic cancer. In addition, the study will evaluate the efficacy of this device in treating pain associated with unresectable pancreatic cancer. Quality of life post-procedure will also be collected.

DETAILED DESCRIPTION:
The NanoKnife, System has been commercially available since 2009, and is FDA-approved to treat soft tissue tumors. The NanoKnife System has received FDA clearance for the surgical ablation of soft tissue. It has not received clearance for the therapy or treatment of any specific disease or condition.

The purpose of this study is to evaluate the short and intermediate term safety of the NanoKnife Irreversible Electroporation System when used off-label to treat unresectable pancreatic cancer. In addition, the study will evaluate the efficacy of this device in treating pain associated with unresectable pancreatic cancer. Quality of life post-procedure will also be collected.

Primary Objective:

• Safety and tolerability of the procedure by monitoring the number of participants with Adverse Events at the following time points: 1, 2, 4, 7, 14, 21 and 30 days and 3, 6, 9, 12, 15, 18, 21, and 24 months post-IRE procedure.

Secondary Objective:

• Pain and Quality of Life outcomes of the patient using Pain Scores on the Visual Analogue Score (VAS) and Quality of Life Scores on the EORTC QLQ-PAN26 and EORTC QLQ-C30 at the following time points: 1, 2, 4, 7, 14, 21 and 30 days and 3, 6, 9, 12, 15, 18, 21, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* > = 18 years of age
* Must be found to have locally advanced unresectable disease following standard chemotherapy ± radiotherapy as demonstrated with either CT/MRI imaging and surgical evaluation, and not have taken any chemotherapy/radiotherapy within 5 weeks of treatment with the NanoKnife IRE System
* Must have an INR < 1.5
* Are willing and able to comply with the protocol requirements
* Are able to comprehend and willing to sign an informed consent form

Exclusion Criteria:

* Creatinine > 2.0 mg/dL
* Any lab value with a grade 3 or 4 toxicity as defined by the CTCAE Version 5.0
* Inability to stop antiplatelet and coumadin therapy for 7 days prior to and 7 days post treatment with the NanoKnife System
* Tumor size not measurable
* Known history of contrast allergy that cannot be medically managed
* Known hypersensitivity to the metal in the electrodes (stainless steel 304L) that cannot be medically managed
* Unable to be treated with a muscle blockade agent (e.g. pancuronium bromide, atracurium, cisatracurium, etc.)
* Women who are pregnant or currently breast feeding
* Women of childbearing potential who are not utilizing an acceptable method of contraception
* Have taken an investigational agent within 30 days of visit 1
* Have implanted cardiac pacemakers or defibrillators
* Have implanted electronic devices or implants with metal parts in the vicinity of a lesion
* Have a history of epilepsy or cardiac arrhythmia (atrial or ventricular fibrillation)
* Have a recent history of myocardial infarction (within the past 2 months)
* Have Q-T intervals greater than 550 ms unless treated with an Accysync Model 72 synchronization system controlling the NanoKnife system's output pulses
* Evidence of distant metastases of stage IV
* Have taken any chemotherapeutic agent within 5 weeks of treatment with the NanoKnife Irreversible Electroporation (IRE) System
* Received non-conventional fractionation schedules, such as stereotactic radiation (5 fractions or less) or received higher than 54 Gray (Gy) delivered conventionally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have unresectable pancreatic cancer following standard chemotherapy with or without radiotherapy will be approached for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Pain | 2 years
  Safety and tolerability of the procedure by monitoring the number of participants with Adverse Events at the following time points: 1, 2, 4, 7, 14, 21 and 30 days and 3, 6, 9, 12, 15, 18, 21, and 24 months post-IRE procedure. The primary endpoint will be the number of Participants with an adverse event related to the IRE treatment and serious or non-serious, at least grade 3, at least possibly related to treatment
  This will be measured by a series of questionnaires on pain scores via Quality of Life scores via the EORTC QLQ-PAN26 and EORTC QLQ-C30. Pain will be measured on a scale from 0-10, with 0 being no pain and 10 being worst pain.
Safety and Pain | 2 years
  Safety and tolerability of the procedure by monitoring the number of participants with Adverse Events at the following time points: 1, 2, 4, 7, 14, 21 and 30 days and 3, 6, 9, 12, 15, 18, 21, and 24 months post-IRE procedure. The primary endpoint will be the number of Participants with an adverse event related to the IRE treatment and serious or non-serious, at least grade 3, at least possibly related to treatment
  This will be measured by a series of questionnaires on pain scores via Visual Analogue Score (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided